CLINICAL TRIAL: NCT04167605
Title: Evaluation of Prognostic Factors: From Breast Cancer to Bone Metastases
Acronym: BC-BOMET
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: BC-BOMET
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Metastatic; Bone Metastases
Keywords: Breast cancer; Bone metastases; SENP1
MeSH Terms: conditions — Breast Neoplasms | interventions — bone metastasis-targeting peptidomimetic-11

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Biological waste material derived from patients undergoing excisional surgery and bone consolidation due to osteolytic bone metastases from breast cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer metastatic to bone: No direct intervention(s) will be administer to the patients. We will use the sample (slides) recovered from the surgery on primary tumor (breast cancer responsible for metastatic disease).
  Interventions: Other: Breast cancer metastatic to bone
- Bone metastasis: No direct intervention(s) will be administer to the patients. Waste material will be analysed for the expression of specific proteins
  Interventions: Other: Bone metastasis

INTERVENTIONS:
Other: Bone metastasis — Collection of waste tissue samples during surgery and immediate immersion of the same in 10% Neutral buffered formalin. The samples will be send to the laboratory where they will be processed (decalcification, inclusion in paraffin, sectioning etc.) for subsequent analyzes.
  Groups: Bone metastasis
Other: Breast cancer metastatic to bone — Patients will be assisted in the recovery of samples (slides) related to surgery on primary tumor (breast cancer responsible for metastatic disease).
  Groups: Breast cancer metastatic to bone

SUMMARY:
Bone metastases represent a frequent complication of some solid tumours, particularly prostate, breast and lung carcinomas. Bone metastases can cause pain and give rise to the so-called "Skeletal-related Events" (SRE) such as pathological fractures and nerve compression. Despite advances in cancer treatment in general, treatment options for bone metastases remain inadequate and generally palliative. It is therefore necessary to identify patients at "high risk" of developing metastases at an early stage of neoplastic disease in order to counteract it. Therefore, the identification of changes in the expression of proteins that could be variously involved in the progression of breast cancer is of primary importance since they could act as prognostic factors and therefore address the therapeutic strategy. The aim of the investigators is to clarify the role of de-regulation of post-translational events (such as SUMOylation) in the progression of breast cancer.

DETAILED DESCRIPTION:
The most serious aspect of neoplastic disease is the spread of cancer cells to secondary sites, often distant from the primary site of growth. Bone is a breeding ground for many types of cancer, especially those derived from breast, prostate and lung. Despite the enormous progress in diagnosis and therapeutic strategies, bone metastases still have a profound impact on quality of life and survival, being often responsible for the outcome of the disease. To improve the outcome of patients with poor prognosis, a deep knowledge of the mechanisms underlying dissemination, colonization and progression of cancer cells in the bone is necessary.

The investigators therefore intend to clarify some pathogenic mechanisms involved in the growth of bone metastases, and to uncover predictive signs that underlie the spread of breast cancer cells to bone.

Primary aim of the investigators is to deepen the role of the de-regulation of post-translational events, such as Small Ubiquitin-like Modifier- (SUMO) SUMO-ylation in the progression of breast cancer. The expression of SENP1 (a member of the SUMO-specific protease family) in bone metastatic and non-metastatic mammary carcinomas will be evaluated. The evaluation of the expression of SENP1 in bone metastases will be finalised to define a possible use as a therapeutic target. SENP1 could be a potential prognostic indicator of the neoplastic progression of breast cancer and a potential therapeutic target, but data on its participation in the process of metastasis to bone are still scarce. Moreover, the investigators try to deepen the knowledge of the interaction between tumour cells and bone microenvironment and the role of immunosurveillance as an important part of the immune response against to neoplastic cells. Finally, the investigators will analyze the role of autophagy and apoptosis in the dissemination and growth of metastases due to the capacity of autophagy to provide energy, nutrients and resistance to anoikis, and to promote the dissemination of cancer cells and metastatic growth.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years) candidates for excisional surgery and bone consolidation due to osteolytic bone metastases from breast cancer.
* Female
* Ability to understand the experimental study and willingness to sign the written consent

Exclusion Criteria:

- Retraction of written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: The population consists of 30 subjects who underwent surgery for bone metastases from breast cancer disease. Within the waste material collected during surgery intervention, it is expected to have 24 samples with an adequate content of metastatic tissue. For 12 of these patients it will be possible to retrieve the sample of the primary breast cancer, and then insert it into the study design. The control group will consist of 12 breast cancer samples that have not shown metastatic development after long follow up and will instead be found in commerce.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-11-12 (Estimated)

PRIMARY OUTCOMES:
SENP1 expression | 6 months
  The expression of SENP1 in bone metastatic mammary carcinomas will be studied. The evaluation of the expression of SENP1 in bone metastases will be finalized to define a possible use as a therapeutic target. The expression of SENP1 in bone metastatic breast carcinoma samples will be compared with the expression of SENP1 in non-metastatic breast cancer (commercial source).

SECONDARY OUTCOMES:
Identification of new predictive molecular markers of breast cancer progression towards an aggressive metastatic state. | 18 months
  Analysis of the expression of proteins involved in the interaction between tumour cells and bone microenvironment, in the immunosurveillance and in the autophagic process in sample of mammary carcinomas that gave rise to bone metastases and in sample of breast cancer without history of bone metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sowder ME, Johnson RW. Bone as a Preferential Site for Metastasis. JBMR Plus. 2019 Jan 15;3(3):e10126. doi: 10.1002/jbm4.10126. eCollection 2019 Mar. PMID 30918918
- [Background] Yeh ET. SUMOylation and De-SUMOylation: wrestling with life's processes. J Biol Chem. 2009 Mar 27;284(13):8223-7. doi: 10.1074/jbc.R800050200. Epub 2008 Nov 13. PMID 19008217
- [Background] Wang Z, Jin J, Zhang J, Wang L, Cao J. Depletion of SENP1 suppresses the proliferation and invasion of triple-negative breast cancer cells. Oncol Rep. 2016 Oct;36(4):2071-8. doi: 10.3892/or.2016.5036. Epub 2016 Aug 24. PMID 27573572
- [Background] Feng Y, Yao Z, Klionsky DJ. How to control self-digestion: transcriptional, post-transcriptional, and post-translational regulation of autophagy. Trends Cell Biol. 2015 Jun;25(6):354-63. doi: 10.1016/j.tcb.2015.02.002. Epub 2015 Mar 8. PMID 25759175
- [Background] Mathew R, Karp CM, Beaudoin B, Vuong N, Chen G, Chen HY, Bray K, Reddy A, Bhanot G, Gelinas C, Dipaola RS, Karantza-Wadsworth V, White E. Autophagy suppresses tumorigenesis through elimination of p62. Cell. 2009 Jun 12;137(6):1062-75. doi: 10.1016/j.cell.2009.03.048. PMID 19524509
- [Background] Moscat J, Diaz-Meco MT. p62 at the crossroads of autophagy, apoptosis, and cancer. Cell. 2009 Jun 12;137(6):1001-4. doi: 10.1016/j.cell.2009.05.023. PMID 19524504